CLINICAL TRIAL: NCT05220124
Title: An Open Label, Randomized Control Study of Probiotics Administration in the Immunotherapy of Urothelial Bladder Carcinoma
Brief Title: A Study of Probiotics Administration in the Immunotherapy of Urothelial Bladder Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Truce-03
Record Dates: First submitted 2022-01-14; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Bladder Urothelial Carcinoma
Keywords: Immunotherapy; Probiotic
MeSH Terms: interventions — Lacteol; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunotherapy with Live Combined (Bifidobacterium,Lactobacillus and Enterococcus Capsules) (Experimental): 420mg Live Combined (Bifidobacterium,Lactobacillus and Enterococcus Capsules) bid for 3-4 treatment cycles,21 days per cycle.
  Interventions: Drug: Live Combined (Bifidobacterium,Lactobacillus and Enterococcus Capsules)
- Immunotherapy without Probiotics (No Intervention): control group, Immunotherapy without Probiotics

INTERVENTIONS:
Drug: Live Combined (Bifidobacterium,Lactobacillus and Enterococcus Capsules) — 420mg Live Combined (Bifidobacterium,Lactobacillus and Enterococcus Capsules) bid for 4 treatment cycles.
  Other Names: Probiotic
  Arms: Immunotherapy with Live Combined (Bifidobacterium,Lactobacillus and Enterococcus Capsules)

SUMMARY:
A study of the efficacy and safety of probiotics in immunotherapy of urothelial carcinoma.

DETAILED DESCRIPTION:
To evaluate the progression free survival of intestinal probiotics in immunotherapy for urothelial carcinoma. Changes in fecal flora abundance before and after treatment were assessed to identify subjects most likely to benefit from enteric probiotics treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with urothelial carcinoma and undergoing immunotherapy ;
2. Age ≥ 18 years;
3. Expected survival time is greater than 12 weeks;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 1 or 2;
5. Organ function level must meet the following requirements:

   Hematological indexes: neutrophil count >= 1.5x10^9/L, platelet count >= 100x10^9/L, hemoglobin >= 9.0 g/dl (can be maintained by symptomatic treatment); Liver function: total bilirubin <=1.5 ULN, alanine aminotransferase and aspartate aminotransferase <=2.5 ULN (can be maintained by symptomatic treatment);
6. The subjects volunteered to join the study, signed informed consent, and had good compliance with follow-up;
7. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Receive live attenuated vaccine within 4 weeks before treatment or during the study period;
2. Active, known or suspected autoimmune diseases;
3. Cannot take orally or are allergic to probiotics ;
4. History of primary immunodeficiency ;
5. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
6. Pregnant or lactating female patients;
7. Untreated acute or chronic active hepatitis B or hepatitis C infection. Under the condition of monitoring the virus copy number of patients receiving antiviral treatment, doctors can judge whether they are in line with the patients' individual conditions;
8. Uncontrolled concurrent diseases, including but not limited to:

HIV infected (HIV antibody positive); Severe infection in active stage or poorly controlled; Evidence of serious or uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [hypertension greater than or equal to conmon terminology criteria for adverse events （CTCAE） grade 2 after drug treatment]); Patients with active bleeding or new thrombotic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 3 years
  Time from randomness to the first occurrence of disease progression or death from any cause.

SECONDARY OUTCOMES:
Duration of Response (DOR) | up to 3 years
  The time from the first judgment of complete response (CR) or partial response (PR) to the discovery of progressive disease （PD）.
Overall Survival (OS) | up to 3 years
  Defined as the number of days from study entry to death. Individuals who are alive at last contact will be censored on the date of last contact.
Serious Adverse Event (SAE) | up to 3 years
  The adverse events that occurred in the study were difficult to manage.
Overall response rate (ORR) | up to 3 years
  defined as the proportion of patients who have a partial or complete response to therapy.
Disease control rate (DCR) | up to 3 years
  The percentage of cases with remission and lesion stability after treatment in the number of evaluable cases.

OTHER OUTCOMES:
16s rDNA sequencing | up to 3 years
  Identify the subgroups that are most likely to benefit from intestinal probiotic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Hu, MD,PhD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China